CLINICAL TRIAL: NCT02860143
Title: Assessment of Ventilation Using Respiratory Volume Monitor During Sedation With Intravenous Propofol as Compared to Capnography in Patients Receiving Intravenous Sedation.
Brief Title: Assessment of Ventilation Using Respiratory Volume Monitor Compared to Capnography During Intravenous Sedation
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bhavani Shankar Kodali, Staff Anesthesiologist, Brigham and Women's Hospital
Other Study IDs: 2014P001522
Record Dates: First submitted 2015-07-28; First posted 2016-08-09 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- studying ventilation during sedation: Comparing ventilation during sedation with capnography

SUMMARY:
A. Determine if Respiratory Volume Monitor (RVM) can be used during procedural sedation to adequately monitor patient's respiratory status as compared to capnograph Aims B. Compare the time of capture of respiratory events (depression, arrest, etc…) on both the RVM and the capnograph C. Compare the incidence of missing or poor quality readings between the RVM and the capnograph D. Compare RR readings between the RVM and the capnograph (during periods with adequate data quality on both devices) E. If RMV can identify respiratory obstruction. Capnography

DETAILED DESCRIPTION:
Rationale for Proposed Research: Continuous respiratory monitoring using the ExSpiron System will be particularly beneficial to patients receiving intravenous propofol breathing spontaneously with natural airway. Assessment and management of respiratory function and early intervention when indicated is a multifaceted, complex task often complicated by the unavailability of a cohesive and continuous monitoring system to guide clinical decisions. The ExSpiron system is designed for these patients and is intended to address some of the limitations of the current generation of hospital monitors and to provide healthcare providers with continuous real-time data regarding the patient's respiratory status. Recent RVM data has shown that stratification of patients based on the MV % of predicted, prior to opioid dosing has made it possible to identify patients who are at risk for further decrease in MV and opioid-induced respiratory depression (OIRD).

1. In the spontaneously breathing, non-ventilated patient, current monitoring devices do not provide continuous, objective non-invasive, continuous real time information of important respiratory parameters such as TV, MV and RR.
2. Current monitoring of non-intubated patients mostly relies on oximetry data, subjective clinical assessment and occasionally EtCO2 measurements. In appropriate clinical settings, the ExSpiron system can provide direct quantitative measure of ventilation parameters for use in clinical assessment and trend prediction as well as response to medications and other interventions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: patient's ≥ 20 years of age receiving intravenous sedation, or intravenous general anesthesia with propofol.

Exclusion Criteria:

Criteria: patients not able to give informed consent, Inability to place the PadSets on the thorax. Existence of an active implanted neurostimulator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients receiving intravenous propofol for sedation, or general anesthesia with natural airway and breathing spontaneously will be recruited and will give written informed consent. The RVM data collection will end when the patient is discharged from the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in minute ventilation, tidal volume, and end-tidal carbon dioxide following propofol | Starting approximately 10 min prior to colonoscopy and continuing until end of colonoscopy (average time: 45-60 minutes)
  Minute ventilation (MV) and tidal volume (TV) measured by the Respiratory Volume Monitor will be reported as percent of baseline established during normal breathing prior to sedation. The percent decrease in MV and TV following propofol will be compared to changes in end-tidal CO2 measured by capnography. The amount of time between propofol doses and changes in MV and TV and EtCO2 will be quantified and compared.

SECONDARY OUTCOMES:
Comparison of Respiratory Rate measurement by Respiratory Volume Monitor and Capnography | Starting approximately 10 min prior to colonoscopy and continuing until end of colonoscopy (average time: 45-60 minutes)
  Respiratory rate measurements from the respiratory volume monitor and capnography will be compared. The percent time that a respiratory rate reading is available will be quantified and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavani Kodali, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No